CLINICAL TRIAL: NCT01604577
Title: Targeting Social Determinants to Improve Chronic Kidney Disease Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kerri Cavanaugh, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120595
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease
Keywords: health literacy; health numeracy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interactive educational intervention (Active Comparator): Physicians will use an interactive educational worksheet during the standard-of-care clinic visit.
  Interventions: Behavioral: interactive educational intervention
- control group (No Intervention): Physicians will conduct the standard-of-care clinic visit as usual.

INTERVENTIONS:
Behavioral: interactive educational intervention — Use of a concise, literacy-sensitive, physician-led, educational interaction with the patient.
  Arms: interactive educational intervention

SUMMARY:
The primary research goals of this application are to characterize social factors including health literacy and numeracy skills of CKD patients and examine associations with knowledge, self-efficacy, self-care behaviors, and clinical outcomes, and to examine the impact of an efficient interactive educational intervention to facilitate patient-provider communication. The investigators will accomplish these goals by executing a cluster-randomized controlled trial and performing detailed analysis of baseline measures. The specific aims of this study are:

Specific Aim 1: Determine the association of social factors with patient kidney knowledge, self-efficacy, participation in self-care behaviors, and clinical outcomes in moderate to advanced CKD.

Hypothesis: In patients with CKD, low health literacy and numeracy is common and associated with older age, non-white race, fewer years of education, lower socioeconomic (income) status, less kidney knowledge, lower self-efficacy of self-care, and less adherence with medication and diet self-care recommendations. Low literacy/numeracy is also associated with higher blood pressures, more proteinuria, and more severe dysfunction of renal clearance.

Specific Aim 2: Evaluate the impact of a tailored literacy-sensitive educational tool used cooperatively by physicians and patients to improve self-care and outcomes in CKD.

Hypothesis: Utilization of a concise literacy-sensitive physician-delivered educational tool will be feasible and associated with higher patient kidney knowledge, self-efficacy of self-care and greater adherence to medication and nutrition recommendations compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care in the Vanderbilt General Nephrology Clinic for at least 1 prior visit past 12 months;
* Serum creatinine available in the medical record in the last 12 months demonstrating Chronic Kidney Disease (eGFR<60mls/min);
* Age 18-80 years;
* English-speaking.

Exclusion Criteria:

* Pre-existing diagnosis of significant dementia or psychosis as determined by primary provider and documented in the medical record;
* Corrected visual Acuity >60/20 using a Rosenbaum Pocket Vision Screen;
* Patient receives dialysis or has a functional kidney transplant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
self-care of Chronic Kidney Disease | baseline and 6 months
  Change from baseline in the following surveys/questionaires at 6 months
  * Morisky 8-Item Survey
  * Frequent Food Questionaire

SECONDARY OUTCOMES:
patient understanding of kidney disease and their disease status | baseline and 6 months
  Change from baseline in the following surveys/questionaires at 6 months
  * Kidney Awareness & Knowledge Survey
  * Perceived Kidney Self-Management Scale
  * Kidney Disease Self-Management Behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Cavanaugh, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States